CLINICAL TRIAL: NCT04117984
Title: Swaziland HIV Incidence Measurement Survey (SHIMS 2, 2016): a Population-based HIV Impact Assessment (PHIA)
Brief Title: Swaziland HIV Incidence Measurement Survey 2
Acronym: SHIMS2
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Ministry of Health, Swaziland (Other Government)
Responsible Party: Principal Investigator, Harriet Nuwagaba-Biribonwoha, Assistant Professor of Epidemiology, Columbia University
Other Study IDs: AAAQ8889; U2GGH001271 (NIH)
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: HIV/AIDS
Keywords: Population-based survey; HIV; Antenatal care; PMTCT; Intimate Partner Violence (IPV); Tuberculosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A repository of dried blood spots and plasma samples will be retained for up to 10 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The second Swaziland HIV Incidence Measurement Survey (SHIMS 2, 2016), is a population based HIV Impact Assessment (PHIA) that will assess the prevalence of key human immunodeficiency virus (HIV)-related health indicators. This is a two-stage cluster sampled cross-sectional survey of 6,417 randomly selected households in Swaziland. Approximately 20,292 eligible persons will be approached (4,664 participants 0-14 years; 12,563 participants 15-49 years; 3,065 participants 50 years and older). Of the sample approached, 15,403 are expected to agree to a blood draw for home-based HIV rapid testing including 3,361 participants 0-14 years; 9,680 participants 15-49 years; and 2,362 participants 50 years and older. SHIMS 2, 2016 will characterize HIV incidence, prevalence, viral load suppression, cluster of differentiation 4 (CD4) T-cell distribution, and risk behaviors in a household-based, nationally-representative sample of the Swazi population and will describe uptake of key HIV prevention, care, and treatment services.

DETAILED DESCRIPTION:
After nearly three decades of Swaziland's national HIV response, a rigorous, population-based measure of the above biological endpoints will provide a valuable follow-up assessment of the impact of the national HIV program. National HIV prevalence and incidence surveys have been carried out in several countries including Uganda (2004), Tanzania (2003), Kenya (2007, 2012), and Swaziland (2011). Specifically in Swaziland, the 2011 SHIMS survey provided critical data on national-level, population-based HIV prevalence, HIV incidence, self-reported antiretroviral therapy (ART) use and viral suppression (VS) among adults 18-49 years. Importantly, SHIMS 2011 lacked data on HIV incidence among participants aged 15-17 years and adults older than 49 years, and HIV prevalence among children 0-14 years. Lack of this vital information limits effective national program planning, resource mobilization, and allocation.

SHIMS 2, 2016 will measure HIV incidence and other HIV-related measures, such as CD4 T-cell count distribution, viral load setpoint (VLS), and prevalence of ARV metabolites and transmitted HIV in Swaziland. SHIMS 2, 2016 will provide an opportunity to characterize the current status of the HIV epidemic and provide greater clarity on the impact of the national HIV program. It will provide important updated information on HIV incidence and uptake of HIV-related services that will allow for measurement of program impact and progress towards 90-90-90 targets. The survey will also estimate the prevalence and distribution of selected behaviors typically associated with HIV acquisition and transmission, for targeted programing in the continued scale-up of HIV services.

SHIMS 2, 2016 will assess the impact of the HIV control efforts in Swaziland, and inform programs moving forward to better tailor the approaches to the most impactful intervention areas and groups that need them. The data will be used to assess country specific HIV indicators, including the impact of the expansion of HIV prevention and treatment programs to facilitate effective monitoring of national HIV programs.

ELIGIBILITY:
Inclusion Criteria:

Participants 18 Years and Older:

1. Resides in selected household or spent the night before the survey there, per above definitions, and
2. Self-reported age 18 years and above, and
3. Ability and willingness to provide written informed consent in English or siSwati

Participants 10-17 Years:

1. Resides in selected household or spent the night before the survey there, per above definitions, and
2. Self-reported age 10-17 years, and
3. Ability and willingness to provide written assent and parent/guardian able and willing to provide written informed consent/permission in English or siSwati, or
4. For children with special circumstances 12-17 years old, ability and willingness to provide written informed consent in English or siSwati

Participants 0-9 Years:

1. Resides in selected household or spent the night before the survey there, per above definitions, and
2. Parent/guardian or child with special circumstances who reports subject's age as 0-9 years, and
3. Parent/guardian/child with special circumstances is able and willing to provide written, informed consent/permission in English or siSwati

Exclusion Criteria:

* Persons who are unable to give consent due to cognitive impairment or intellectual disability will not be eligible to participate. (Individuals with other disabilities who are otherwise able to give written informed consent, mark, or thumb print will be offered survey participation.)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sampling frame will be comprised of all households in the country, based on the 2007 Population and Housing Census of Swaziland. The sampling frame consists of 2,064 EAs, containing 212,195 households and 1,005,206 persons, with an average number of 105 households per EA.
Sampling Method: Probability Sample
Enrollment: 15429 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
HIV incident rate among adults 15 years and older | 1 year
  The survey will allow calculation of a national HIV incidence estimate using HIV-1 Limiting Antigen (LAg)-Avidity Enzyme Immunoassay
Sub-national prevalence of suppressed HIV viral load (<1,000 copies/mL) among adults 15 and older | 1 year
  Viral load (VL) (viral copies/mL) of HIV-infected participants will be measured using Abbott, Roche, or similar platform
HIV prevalence of children ages 0-14 | 1 year
  A representation of the child population will be sampled

SECONDARY OUTCOMES:
HIV Prevalence in 2016 among adults 15 years and older | 1 year
  The entire adult population will be sampled
HIV incidence estimates among young women aged 18-24 in 2011 versus 2016 | 1 year
  The incidence estimates measured in 2016 will be compared to the previous survey incidence estimates in 2011
Incidents of HIV infection among adults from risky behaviors | 1 year
  Questionnaire indicators will be used for this measure, specifically questions on sexual behavior and other risky behaviors
Mean population viral load among adults living with HIV | 1 year
  Viral load of HIV-infected participants will be measured using Abbott, Roche, or a similar platform
Prevalence of adult viral suppression in 2011 versus 2016 | 1 year
  The viral load suppression measured in 2016 will be compared to the previous survey in 2011, national and regional
CD4+ count distribution of adults living with HIV | 1 year
  The total population of HIV positive adults will be sampled, national
Enrollment rate in HIV care among adults with prevalent HIV infection | 1 year
  Questionnaire indicators will be used for this measure
Prevalence of antiretroviral therapy (ART) use among adults and children with prevalent HIV infection | 1 year
  Questionnaire indicators will be used for this measure
Uptake of HIV testing and ART use among women recently pregnant or breastfeeding | 1 year
  Questionnaire indicators will be used for this measure
Prevalence of transmitted antiretroviral (ARV) drug resistance (DR) among adults and children with recent HIV infection | 1 year
  The sub population of HIV infected individuals will be sampled
Prevalence of viral suppression among adults and children on ART | 1 year
  Questionnaire indicators will be used for this measure
Incidence of reported sexual behavior associated with HIV transmission risk among adults | 1 year
  Questionnaire indicators will be used for this measure, specifically questions on sexual behavior and other risky behaviors
Percentage of prior testing and knowledge of HIV status among adults | 1 year
  Questionnaire indicators will be used for this measure
Prevalence of male circumcision among men 15 years and older and among male children | 1 year
  Questionnaire indicators will be used for this measure
Uptake of tuberculosis services among adults | 1 year
  Questionnaire indicators will be used for this measure
Acceptability rate of early ART use among adults who test HIV sero-positive and self report as not currently on ART | 1 year
  Questionnaire indicators will be used for this measure
Prevalence of HIV infection among children | 1 year
  Questionnaire indicators will be used for this measure
Enrollment rate in HIV care among HIV-infected children | 1 year
  Questionnaire indicators will be used for this measure
CD4+ count distribution of children living with HIV | 1 year
  The total population of HIV positive children will be sampled, national
Prevalence of sub-national viral suppression among children living with HIV | 1 year
  Viral load of HIV-infected participants will be measured using Abbott, Roche, or similar platform
Prevalence of sexual behavior and debut associated with HIV transmission risk among participants aged 10-14 years | 1 year
  Questionnaire indicators will be used for this measure, specifically questions on sexual behavior and other risky behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Justman, MD, Study Director — Columbia University; David Hoos, MD, Study Director — Columbia University; Harriet Nuwagaba-Biribonwoha, MD, Principal Investigator — Columbia University
Locations (1):
- ICAP at Columbia University, Mbabane, Eswatini

IPD SHARING:
Plan to Share IPD: Yes
Data will be anonymised, and will be part of a public release dataset released approximately 12 months after data collection ceases via a SHIMS website.
Time Frame: Approximately 12 months after data collection ceases.
Access Criteria: Public release dataset.

REFERENCES:
- [Background] West CA, Chang GC, W Currie D, Bray R, Kinchen S, Behel S, McCullough-Sanden R, Low A, Bissek A, Shang JD, Ndongmo CB, Dokubo EK, Balachandra S, Lobognon LR, Dube L, Nuwagaba-Biribonwoha H, Li M, Pasipamire M, Getaneh Y, Lulseged S, Eshetu F, Kingwara L, Zielinski-Gutierrez E, Tlhomola M, Ramphalla P, Kalua T, F Auld A, B Williams D, Remera E, Rwibasira GN, Mugisha V, Malamba SS, Mushi J, Jalloh MF, Mgomella GS, Kirungi WL, Biraro S, C Awor A, Barradas DT, Mugurungi O, H Rogers J, Bronson M, M Bodika S, Ajiboye A, Gaffga N, Moore C, Patel HK, C Voetsch A. Unawareness of HIV Infection Among Men Aged 15-59 Years in 13 Sub-Saharan African Countries: Findings From the Population-Based HIV Impact Assessments, 2015-2019. J Acquir Immune Defic Syndr. 2021 Aug 1;87(Suppl 1):S97-S106. doi: 10.1097/QAI.0000000000002708. PMID 34166316
- [Background] Voetsch AC, Duong YT, Stupp P, Saito S, McCracken S, Dobbs T, Winterhalter FS, Williams DB, Mengistu A, Mugurungi O, Chikwanda P, Musuka G, Ndongmo CB, Dlamini S, Nuwagaba-Biribonwoha H, Pasipamire M, Tegbaru B, Eshetu F, Biraro S, Ward J, Aibo D, Kabala A, Mgomella GS, Malewo O, Mushi J, Payne D, Mengistu Y, Asiimwe F, Shang JD, Dokubo EK, Eno LT, Zoung-Kanyi Bissek AC, Kingwara L, Junghae M, Kiiru JN, Mwesigwa RCN, Balachandra S, Lobognon R, Kampira E, Detorio M, Yufenyuy EL, Brown K, Patel HK, Parekh BS. HIV-1 Recent Infection Testing Algorithm With Antiretroviral Drug Detection to Improve Accuracy of Incidence Estimates. J Acquir Immune Defic Syndr. 2021 Aug 1;87(Suppl 1):S73-S80. doi: 10.1097/QAI.0000000000002707. PMID 34166315
- [Background] Reid G, Voetsch AC, Stupp P, McCracken S, Kalton G, Dlamini S, McOllogi Juma J, Kalua T, Kirungi W, Koto M, Mugurungi O, Mulenga L, Mutenda N, Marum L, Saito S. Improving Sampling Efficiency for Determining Pediatric HIV Prevalence in National Surveys: Evidence From 8 Sub-Saharan African Countries. J Acquir Immune Defic Syndr. 2021 Aug 1;87(Suppl 1):S43-S51. doi: 10.1097/QAI.0000000000002704. PMID 34166312
- [Background] Porter L, Bello G, Nkambule R, Justman J. HIV General Population Surveys: Shedding Light on the Status of HIV Epidemics and Informing Future Actions. J Acquir Immune Defic Syndr. 2021 Aug 1;87(Suppl 1):S2-S5. doi: 10.1097/QAI.0000000000002701. PMID 34166307
- [Background] Patel HK, Duong YT, Birhanu S, Dobbs T, Lupoli K, Moore C, Detorio M, Sleeman K, Manjengwa J, Wray-Gordon F, Yavo D, Jackson K, Domaoal RA, Yufenyuy EL, Vedapuri S, Ndongmo CB, Ogollah FM, Dzinamarira T, Rubinstein P, Sachathep KK, Metz M, Longwe H, Saito S, Brown K, Voetsch AC, Parekh BS. A Comprehensive Approach to Assuring Quality of Laboratory Testing in HIV Surveys: Lessons Learned From the Population-Based HIV Impact Assessment Project. J Acquir Immune Defic Syndr. 2021 Aug 1;87(Suppl 1):S17-S27. doi: 10.1097/QAI.0000000000002702. PMID 34166309
- [Background] Hines JZ, Sachathep K, Pals S, Davis SM, Toledo C, Bronson M, Parekh B, Carrasco M, Xaba S, Mandisarisa J, Kamobyi R, Chituwo O, Kirungi WL, Alamo S, Kabuye G, Awor AC, Mmbando S, Simbeye D, Aupokolo MA, Zemburuka B, Nyirenda R, Msungama W, Tarumbiswa T, Manda R, Nuwagaba-Biribonwoha H, Kiggundu V, Thomas AG, Watts H, Voetsch AC, Williams DB. HIV Incidence by Male Circumcision Status From the Population-Based HIV Impact Assessment Surveys-Eight Sub-Saharan African Countries, 2015-2017. J Acquir Immune Defic Syndr. 2021 Aug 1;87(Suppl 1):S89-S96. doi: 10.1097/QAI.0000000000002658. PMID 33765683
- [Background] Bray R, Palma AM, Philip NM, Brown K, Levin B, Thompson JLPS, Ginindza C, Mulenga LB. Is Interview Length Associated With Blood Test Participation? Evidence From Three Population-Based HIV Impact Assessment Surveys Conducted From 2016 to 2017. J Acquir Immune Defic Syndr. 2021 Aug 1;87(Suppl 1):S57-S66. doi: 10.1097/QAI.0000000000002705. PMID 34166313
- [Background] Jonnalagadda S, Yuengling K, Abrams E, Stupp P, Voetsch A, Patel M, Minisi Z, Eliya M, Hamunime N, Rwebembera A, Kirungi W, Mulenga L, Mushavi A, Ryan C, Ts'oeu M, Kim E, Dziuban EJ, Hageman K, Galbraith J, Mweebo K, Mwila A, Gonese E, Patel H, Modi S, Saito S. Survival and HIV-Free Survival Among Children Aged </=3 Years - Eight Sub-Saharan African Countries, 2015-2017. MMWR Morb Mortal Wkly Rep. 2020 May 15;69(19):582-586. doi: 10.15585/mmwr.mm6919a3. PMID 32407305
- [Background] Saito S, Chung H, Mahy M, Radin AK, Jonnalagadda S, Hakim A, Awor AC, Mwila A, Gonese E, Wadonda-Kabondo N, Rwehumbiza P, Ao T, Kim EJ, Frederix K, Nuwagaba-Biribonwoha H, Musuka G, Mugurungi O, Mushii J, Mnisi Z, Munthali G, Jahn A, Kirungi WL, Sivile S, Abrams EJ. Pediatric HIV Treatment Gaps in 7 East and Southern African Countries: Examination of Modeled, Survey, and Routine Program Data. J Acquir Immune Defic Syndr. 2018 Aug 15;78 Suppl 2:S134-S141. doi: 10.1097/QAI.0000000000001739. PMID 29994836
- [Background] Justman JE, Mugurungi O, El-Sadr WM. HIV Population Surveys - Bringing Precision to the Global Response. N Engl J Med. 2018 May 17;378(20):1859-1861. doi: 10.1056/NEJMp1801934. No abstract available. PMID 29768142
- [Background] Dwyer-Lindgren L, Cork MA, Sligar A, Steuben KM, Wilson KF, Provost NR, Mayala BK, VanderHeide JD, Collison ML, Hall JB, Biehl MH, Carter A, Frank T, Douwes-Schultz D, Burstein R, Casey DC, Deshpande A, Earl L, El Bcheraoui C, Farag TH, Henry NJ, Kinyoki D, Marczak LB, Nixon MR, Osgood-Zimmerman A, Pigott D, Reiner RC Jr, Ross JM, Schaeffer LE, Smith DL, Davis Weaver N, Wiens KE, Eaton JW, Justman JE, Opio A, Sartorius B, Tanser F, Wabiri N, Piot P, Murray CJL, Hay SI. Mapping HIV prevalence in sub-Saharan Africa between 2000 and 2017. Nature. 2019 Jun;570(7760):189-193. doi: 10.1038/s41586-019-1200-9. Epub 2019 May 15. PMID 31092927